CLINICAL TRIAL: NCT00762099
Title: The Short and Long Term Effects of Perioperative Pregabalin Use on Functional Rehabilitation, Pain Outcomes and Anxiety Following Total Hip Arthroplasty: A Randomized, Double-Blind, Placebo-Controlled Trial.
Brief Title: Perioperative Pregabalin Use, Rehabilitation, Pain Outcomes and Anxiety Following Hip Surgery
Acronym: RCT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Dr. Hance Clarke, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2008-PFE-01
Record Dates: First submitted 2008-09-29; First posted 2008-09-30 (Estimated); Last update posted 2011-04-08 (Estimated); Status verified 2011-04

CONDITIONS: Anxiety
Keywords: Arthroplasty, Hip; Hip replacement; Pain Management; Functional Rehabilitation; Anxiety; Perioperative; Pregabalin; Arthroplasty
MeSH Terms: conditions — Anxiety Disorders; Agnosia | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Pregabalin Group
  Interventions: Drug: Pregabalin
- 2 (Placebo Comparator): Placebo group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregabalin — Pre-operative dose 150 mg Post-operative dose 75 mg BID
  Other Names: Lyrica
  Arms: 1
Drug: Placebo — Placebo/sugar tabs will look identical to active drug.
  Arms: 2

SUMMARY:
Pain prior to surgery is of particular concern in patients undergoing total hip arthroplasty (THA) since it is the most important predictor of pain and poor function 2-3 years after surgery. Previous studies have investigated various treatments for managing pain during and after surgery. However, no study has investigated the short and long term effects of pregabalin in terms of functional rehabilitation, pain outcome and anxiety following total hip arthroplasty. Therefore, the aim of the present study is determine if the following: (1) if perioperative pregabalin administration positively influence early rehabilitation and recovery of physical function and to determine if these effects maintained at 6 weeks and 3 months post surgery. (2) To determine if perioperative pregabalin administration reduce postoperative movement evoked pain associated with rehabilitation and if these effects also maintained at 6 weeks and 3 months post surgery.

DETAILED DESCRIPTION:
INTRODUCTION. Participants are being asked to consider taking part in this research study if they are scheduled for total hip surgery. In this study we will compare the effect of a pain medication known as Pregabalin compared to placebo on rehabilitation and recovery of physical function and pain associated with rehabilitation. We will monitor patient progress in hospital and follow-up participants at 6 weeks and 3 months post surgery.

At the Holland Orthopedic and Arthritic Centre we use different methods to control postoperative pain. Postoperative pain relief is usually controlled with morphine using a pump that participants can control themselves, sometimes called "PCA" (Patient Controlled Analgesia). Participants also receive a combination of tablets like an anti-inflammatory (Celecoxib), and opioids (strong pain killers), to get the best pain relief possible with the fewest side effects. Anti-Inflammatories are a type of pain medicine that reduces swelling (inflammation). We would like to see compare the recovery profile of participants who receive in their pain management plan, the addition of Pregabalin with those who receive placebo.

WHY IS THIS STUDY BEING DONE? Pregabalin has recently been shown to reduce the amount of morphine participants use after surgery and enhance rehabilitation in some orthopedic participants. This study will examine whether Pregabalin added to a patient's pain management plan will help them rehabilitate more effectively and with less pain.

Part of this research will involve the collection of information from study participants that describes any pain or discomfort that they experience before and after surgery. After surgery, participants will be asked about how much pain they have by the nursing staff. In order to address these issues, they are asked to provide the following information at various intervals during their hospital stay:

1. Pain intensity - using a Numeric Rating Scale (NRS) where 0=no pain and 10=Terrible Pain will be recorded three times daily during your hospital stay. Participants will also be asked to rate their pain after several rehabilitation measures on Postoperative days 1 to 4.
2. Participants will also be asked if they are feeling nauseated, feel like vomiting, or feel drowsy.

After Total Hip Arthroplasty, it is important that all patients receive a standardized rehabilitation protocol. At the Holland Orthopedic and Arthritic Centre, the Primary Hip Replacement Care Pathway is accompanied by a standardized rehabilitation treatment protocol. While patients are in hospital, they will meet a physiotherapist who will put them through a series of hip exercises. The physiotherapist will record how much movement they can perform with their hip every day that they are in hospital.

On postoperative day 2 and day 4 study participants will, in addition to their daily hip exercises, be asked to perform a walking test to the best of ability. Participants will be timed, the physiotherapist will ask the participant to stand from a chair and walk 3 meters at a comfortable safe pace. Participants will then turn and walk back to the chair, and then sit down. In order that participants are familiar with that test we will perform that exercise before their operation so that we can obtain a baseline score. At the completion of the walking test, participants will also be asked to provide a final pain assessment of how painful the walking test was. On postoperative day 4, and at 6 weeks and at 3 months participants will be asked to perform some other rehabilitation measures. One will be a timed six minute walk test (only at 6 weeks and 3 months), that means we will measure how far they can walk in 6 minutes. The other measure will be one requiring participants to walk up stairs, they will have a good understanding of the above tests because they will have performed these tests prior to surgery.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent, American Society of Anesthesiologists physical status I-III, VAS > 5, age18-75 years, male or female, scheduled for THA.

Exclusion Criteria:

Patients will not be enrolled in this study for the following reasons:

* Patients not providing informed consent.
* Known allergy to any of the medications being used.
* History of drug or alcohol abuse.
* Patients with chronic pain on slow-release preparations of opioid.
* Patients with Rheumatoid Arthritis.
* Patients with psychiatric disorders.
* Patients unable or unwilling to use Patient Controlled Analgesia. (PCA)
* Diabetic patients or those with impaired renal function (Creatinine >106).
* Obese patients (i.e. BMI > 40).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2009-05; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Physical function 6 weeks and 3-months post-total hip arthroplasty | Up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Colin McCartney, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Holland Orthopaedic and Arthritic Centre, Toronto, Ontario, Canada